CLINICAL TRIAL: NCT02621944
Title: Melatonin as a Neuroprotective Therapy in Neonates With HIE Undergoing Hypothermia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201500886
Record Dates: First submitted 2015-10-19; First posted 2015-12-04 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hypoxic Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Melatonin; Magnetic Resonance Spectroscopy; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Participants 1-10 (Experimental): This group will receive a 0.5 mg/kg enteral dose of Melatonin. The first dose will be administered via enteral route within 12 hours of life with a target of 6 hours of life.
  The melatonin will be administered as a single dose for the first 5 participants in allowing the investigators to determine if the dosing frequency has the potential to decrease in the elimination with hypothermia. The next 5 subjects who will receive multiple doses if there are not any safety concerns.
  Additionally, the participants will have the following test performed: Magnetic Resonance Imaging (MRI), Neurological Outcome Assessment, Pharmacokinetics, and safety monitoring.
  Interventions: Drug: Melatonin; Other: Magnetic Resonance Imaging; Other: Pharmacokinetics; Behavioral: Neurological Outcome Assessment
- Participants 11-20 (Experimental): This group will the Melatonin dose of 3 mg/kg enteral, only if the group Participants 1-10 has meet the safety goals. The first dose will be administered via enteral route within 12 hours of life with a target of 6 hours of life.
  The melatonin will be administered as a single dose for the first 5 participants in allowing the investigators to determine if the dosing frequency has the potential to decrease in the elimination with hypothermia. The next 5 subjects who will receive multiple doses if there are not any safety concerns.
  Additionally, the participants will have the following test performed: Magnetic Resonance Imaging (MRI), Neurological Outcome Assessment, Pharmacokinetics, and safety monitoring.
  Interventions: Drug: Melatonin; Other: Magnetic Resonance Imaging; Other: Pharmacokinetics; Behavioral: Neurological Outcome Assessment
- Participants 21-30 (Experimental): This group will receive Melatonin dose of 5 mg/kg enterally, only if the group Participants 11-20 has meet the safety goals. The first dose will be administered via enteral route within 12 hours of life with a target of 6 hours of life.
  The melatonin will be administered as a single dose for the first 5 participants in allowing the investigators to determine if the dosing frequency has the potential to decrease in the elimination with hypothermia. The next 5 subjects who will receive multiple doses if there are not any safety concerns.
  Additionally, the participants will have the following test performed: Magnetic Resonance Imaging (MRI), Neurological Outcome Assessment, Pharmacokinetics, and safety monitoring.
  Interventions: Drug: Melatonin; Other: Magnetic Resonance Imaging; Other: Pharmacokinetics; Behavioral: Neurological Outcome Assessment

INTERVENTIONS:
Drug: Melatonin — Participants 1-10 will receive a 0.5 mg/kg enteral dose of Melatonin. Participants 11-20 will receive Melatonin dose of 3 mg/kg enteral. Participants 21-30 will receive Melatonin dose of 5 mg/kg enterally.
Other: Magnetic Resonance Imaging — All participants will receive an MRI between 7-12 days of age.
  Other Names: MRI
Other: Pharmacokinetics — All participants will receive pharmacokinetics to test the amount of melatonin in the blood.
Behavioral: Neurological Outcome Assessment — All participants will receive the Bayley-III Scores and Subsets for neurological outcome assessments.

SUMMARY:
Hypoxic-Ischemic Encephalopathy (HIE) occurs in 20 per 1000 births. Only 47% of neonates treated with the state of the art therapy (induced systemic hypothermia) have normal outcomes. Therefore, other promising therapies that potentially work in synergy with hypothermia to improve neurologic outcomes need to be tested. One potential agent is melatonin. Melatonin is a naturally occurring substance produced mainly from the pineal gland. Melatonin is widely known for its role in regulating the circadian rhythm, but it has many other effects that may benefit infants with HI injury. Melatonin serves as a free radical scavenger, decreases inflammatory cytokines, and stimulates anti-oxidant enzymes. Therefore, melatonin may interrupt several key components in the pathophysiology of HIE, in turn minimizing cell death and improving outcomes. The research study will evaluate the neuroprotective properties and appropriate dose of Melatonin to give to infants undergoing therapeutic hypothermia for hypoxic ischemic encephalopathy.

DETAILED DESCRIPTION:
Thirty subjects will be enrolled in a dose escalation study. Subjects 1-10 will receive melatonin (0.5 mg/kg). If that dose proves to be safe, subjects 11-20 will receive an increased dose of melatonin (3 mg/kg). Subjects 21-30 will receive a dose increased to the targeted projected therapeutic dose (5 mg/kg).

The serum concentration of melatonin and capture adverse event reports during this dose escalation study in neonates undergoing hypothermia and the long-term safety and potential efficacy via developmental follow-up performed at 18-22 months of age. In addition, this study will determine the effect of melatonin on the inflammatory cascade, oxidative stress, free radical production, and serum biomarkers of brain injury in neonates undergoing hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* Eligible infants are >36 0/7th weeks gestation,
* pH (cord or neonatal) <7.0,
* base deficit >16 mEq/L,
* no available blood gas,
* a cord blood/first hour of life blood gas with pH > 7.0 and < 7.15,
* base deficit between 10 and 15.9 mEq/L,
* infants must have a history of an acute perinatal event,
* either a 10-minute Apgar < 5 or a continued need for ventilation,
* All infants must have signs of encephalopathy within 6 hours of age using the modified Sarnat scoring system,
* neonates cooled within 6 hours of birth will be included in the study.

Exclusion Criteria:

* suspected inborn errors of metabolism (elevated ammonia) and hypoglycemia,
* clinical signs and symptoms consistent with meningitis detected upon sepsis evaluation,
* a diagnosis of congenital abdominal surgical problems along with multiple congenital anomalies and/or chromosomal abnormalities.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2016-11; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To identify the maximum tolerated dose of Melatonin | Changes in Baseline to day 3
  The maximum tolerated dose (MTD) is defined as the highest dose level without adverse events in no more than 1 out of 6 patients
Bayley-III Index Scores (Cognitive, Language, and Motor) will be used for neurological outcome assessment | Approximately 18 - 20 Months
  All raw scores will be transformed into norm-referenced standard scores (scale mean = 100 with s.d. = 15) using the Bayley-III scoring software published with the test. To dichotomize "good" and "poor" outcomes for statistical analysis, standardized scores that are at or greater than one standard deviation below the normative sample mean published with the test (i.e., standard scores < 85) will be classified as "poor outcome" while higher scores will be classified as "good outcome".
Peak Plasma Concentration (Cmax) of Melatonin 0.5 mg/kg. | 0 (baseline), 3, 5, 6, 12, 24, 48, 96 hours and day 14 (one sample)
  HPLC-ESI/MS/MS will be used to measure melatonin concentrations in the serum samples. The two-way ANOVA (treatments are dose level and timepoint) framework for testing. Testing will be done using a likelihood ratio test, either using large-sample theory approximation or using bootstrap.
Number of participants with treatment-related adverse events as assessed by MedDRA ??? This is something the PI/Team needs to agree on which one to use. | Baseline ongoing to Day 14
  Incidence/Grade of Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), laboratory abnormalities Percentage and number of subjects who discontinued for adverse event
Peak Plasma Concentration (Cmax) of Melatonin 3 mg/kg. | 0 (baseline), 3, 5, 6, 12, 24, 48, 96 hours and day 14 (one sample)
  HPLC-ESI/MS/MS will be used to measure melatonin concentrations in the serum. The two-way ANOVA (treatments are dose level and timepoint) framework for testing. Testing will be done using a likelihood ratio test, either using large-sample theory approximation or using bootstrap.
Peak Plasma Concentration (Cmax) of Melatonin 5 mg/kg. | 0 (baseline), 3, 5, 6, 12, 24, 48, 96 hours and day 14 (one sample)
  HPLC-ESI/MS/MS will be used to measure melatonin concentrations in the serum samples. The two-way ANOVA (treatments are dose level and timepoint) framework for testing. Testing will be done using a likelihood ratio test, either using large-sample theory approximation or using bootstrap.

SECONDARY OUTCOMES:
Bayley-III Index Scores Subscales (Receptive and Expressive Language, Fine and Gross Motor) will be used for neurological outcome assessment | Approximately 18 - 20 Months
  The four performance-based subscales of the Bayley-III Index Scores (Receptive and Expressive Language, Fine and Gross Motor) and two parent-reported scales (Social-Emotional and Adaptive Behavior) will be collected. All raw scores will be transformed into norm-referenced standard scores (scale mean = 100 with s.d. = 15) using the Bayley-III scoring software published with the test. To dichotomize "good" and "poor" outcomes for statistical analysis, standardized scores that are at or greater than one standard deviation below the normative sample mean published with the test (i.e., standard scores < 85) will be classified as "poor outcome" while higher scores will be classified as "good outcome".
Evaluation of The Impact of Melatonin using Magnetic Resonance Image (MRI) | Approximately 7 - 12 days
  The MRI study scores of neonates treated with hypothermia plus melatonin will be compared with historical controls that have matched Sarnat exams (exam of HIE severity at the time of admission).

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Weiss, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Florida Hospital for Children, Orlando, Florida